CLINICAL TRIAL: NCT03998059
Title: Evaluation of Immune Status Before and After Splenectomy in Immune Thrombocytopenia Patients
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: KT2018087
Record Dates: First submitted 2019-06-13; First posted 2019-06-25 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-08

CONDITIONS: Thrombocytopenia; Splenectomy
Keywords: Thrombocytopenia; splenectomy
MeSH Terms: conditions — Thrombocytopenia | interventions — Splenectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 30 immune thrombocytopenia(ITP) patients: A total of 30 cases. The investigators plan to take 20ml of peripheral blood (PB) of these 30 ITP patients at 6 time points, including 1 day before surgery, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery
  Interventions: Procedure: splenectomy
- 20 normal controls: A total of 20 cases.18 age- and gender- matched healthy donor will also be enrolled as controls and taken 20ml of peripheral blood.
- Spleens of the 30 cases patients(ITP): These 30 ITP patients agree to have splenectomy.The investigators will take a small amount of spleen tissue during surgery.
- Spleens of the 10 cases patients(normal controls): The investigators also plan to take splenic tissue from 10 patients who have splenectomy due to hereditary spherocytosis or trauma.

INTERVENTIONS:
Procedure: splenectomy — These patients should fail to have sustained response to multiple first- and second-line treatments of ITP and agree to have splenectomy.Before splenectomy, these patients will be reassessed and still diagnosed with ITP.Their platelet level will be raised to a safe state before surgery, and the laparoscopic splenectomy will be performed in Tianjin People's Hospital.
  Groups: 30 immune thrombocytopenia(ITP) patients

SUMMARY:
Evaluation of immune status before and after splenectomy in immune thrombocytopenia patients.

DETAILED DESCRIPTION:
A total of 30 ITP patients will be enrolled in the study. These patients should fail to have sustained response to multiple first- and second-line treatments of ITP and agree to have splenectomy. Before splenectomy, these patients will be reassessed and still diagnosed with ITP.Their platelet level will be raised to a safe state before surgery, and the laparoscopic splenectomy will be performed in Tianjin People's Hospital. The investigators plan to take 20ml of peripheral blood (PB) of these patients at 6 time points, including 1 day before surgery, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery, and take a small amount of spleen tissue during surgery.

18 age- and gender- matched healthy donor will also be enrolled as controls and taken 20ml of peripheral blood. The investigators also plan to take splenic tissue from 10 patients who have splenectomy due to Hereditary spherocytosis or trauma.

And then the investigators will do the experiments step by step. 1, Isolation of peripheral blood and splenic mononuclear cells;2, Detection of the percentage of cell population;3, Activation and proliferation of B lymphocyte; 4, Activation and proliferation of T lymphocyte;5,Apoptosis of platelets by cytotoxic T cells;6,Phagocytosis of platelets by macrophages in spleen;7,Enzyme-linked immunosorbent assay (ELISA) for cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years old, male or female;
* Conform to the diagnostic criteria of immune Thrombocytopenia (ITP)
* Needed splenectomy;
* People who are willing to sign the informed consent voluntarily and follow the research program.

Exclusion Criteria:

* Secondary thrombocytopenic purpura;
* Patients with poor compliance;
* Researchers believe that patients should not participate in the test of any other condition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The ITP patients who are eligible for inclusion, but not eligible for exclusion, will be included in the clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2025-07-23 (Estimated)

PRIMARY OUTCOMES:
Changes of the percentage of cell population | 1 year
  To assess the changes of the percentage of B cell subsets，regulatory B cells（Breg），regulatory T cells (Treg)，supressor T cells（Ts），monocyte Fc receptor（FCR）I/II, FCRIII and FCRIIb, helper T cells（Th）subsets and the functionally-polarized CD4+ T cell subsets in peripheral blood mononuclear cells（PBMCs）at 6 time points, including 1 day before surgery, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery, and to compare with the healthy controls.
Changes of activation and proliferation of B and T lymphocyte, apoptosis of platelets by cytotoxic T cells(CTLs) | 1 year
  To assess the changes of activation and proliferation of B and T lymphocyte, apoptosis of platelets by cytotoxic T cells(CTLs) in peripheral blood mononuclear cells（PBMCs）at 6 time points, including 1 day before surgery, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery, and to compare with the healthy controls.
Changes of cytokines in the cell culture supernatants and plasma | 1 year
  To assess the changes of cytokines in the cell culture supernatants and plasma at 6 time points, including 1 day before surgery, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery, and to compare with the healthy controls.

SECONDARY OUTCOMES:
Changes of phagocytosis of platelets by macrophages in itp patients spleen and the normal spleen controls. | The day of the splenectomy
  To assess the changes of phagocytosis of platelets by macrophages in itp patients spleen and the normal spleen controls.
Changes of the percentage of cell population, activation and proliferation of B and T lymphocyte, apoptosis of platelets by cytotoxic T cells(CTLs) in itp patients spleen and the normal spleen controls. | The day of the splenectomy
  To assess the changes of the percentage of B cell subsets，regulatory B cells（Breg），regulatory T cells (Treg)，supressor T cells（Ts），monocyte Fc receptor（FCR）I/II, FCRIII and FCRIIb, helper T cells（Th）subsets ,the functionally-polarized CD4+ T cell subsets, activation and proliferation of B and T lymphocyte, apoptosis of platelets by cytotoxic T cells(CTLs) in itp patients spleen and the normal spleen controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Yunfei Chen, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olsson B, Ridell B, Jernas M, Wadenvik H. Increased number of B-cells in the red pulp of the spleen in ITP. Ann Hematol. 2012 Feb;91(2):271-7. doi: 10.1007/s00277-011-1292-2. Epub 2011 Jul 23. PMID 21785982
- [Background] Kuwana M, Okazaki Y, Kaburaki J, Kawakami Y, Ikeda Y. Spleen is a primary site for activation of platelet-reactive T and B cells in patients with immune thrombocytopenic purpura. J Immunol. 2002 Apr 1;168(7):3675-82. doi: 10.4049/jimmunol.168.7.3675. PMID 11907134
- [Background] Zhang F, Chu X, Wang L, Zhu Y, Li L, Ma D, Peng J, Hou M. Cell-mediated lysis of autologous platelets in chronic idiopathic thrombocytopenic purpura. Eur J Haematol. 2006 May;76(5):427-31. doi: 10.1111/j.1600-0609.2005.00622.x. Epub 2006 Feb 15. PMID 16480433
- [Background] Liu B, Zhao H, Poon MC, Han Z, Gu D, Xu M, Jia H, Yang R, Han ZC. Abnormality of CD4(+)CD25(+) regulatory T cells in idiopathic thrombocytopenic purpura. Eur J Haematol. 2007 Feb;78(2):139-43. doi: 10.1111/j.1600-0609.2006.00780.x. PMID 17328716
- [Background] Ling Y, Cao X, Yu Z, Ruan C. Circulating dendritic cells subsets and CD4+Foxp3+ regulatory T cells in adult patients with chronic ITP before and after treatment with high-dose dexamethasome. Eur J Haematol. 2007 Oct;79(4):310-6. doi: 10.1111/j.1600-0609.2007.00917.x. Epub 2007 Aug 10. PMID 17692100
- [Background] Olsson B, Ridell B, Carlsson L, Jacobsson S, Wadenvik H. Recruitment of T cells into bone marrow of ITP patients possibly due to elevated expression of VLA-4 and CX3CR1. Blood. 2008 Aug 15;112(4):1078-84. doi: 10.1182/blood-2008-02-139402. Epub 2008 Jun 2. PMID 18519809
- [Background] McMillan R, Wang L, Tani P. Prospective evaluation of the immunobead assay for the diagnosis of adult chronic immune thrombocytopenic purpura (ITP). J Thromb Haemost. 2003 Mar;1(3):485-91. doi: 10.1046/j.1538-7836.2003.00091.x. PMID 12871454
- [Background] Yu J, Heck S, Patel V, Levan J, Yu Y, Bussel JB, Yazdanbakhsh K. Defective circulating CD25 regulatory T cells in patients with chronic immune thrombocytopenic purpura. Blood. 2008 Aug 15;112(4):1325-8. doi: 10.1182/blood-2008-01-135335. Epub 2008 Apr 17. PMID 18420827